CLINICAL TRIAL: NCT05666180
Title: Impact of Complicated and Uncomplicated Traumatic Dental Injuries on Oral Health-Related Quality of Life of a Group of Preschool Children and Their Families: Cross-sectional Study
Brief Title: Impact of Complicated and Uncomplicated Traumatic Dental Injuries on Oral Health-related Quality of Life of a Group of Preschool Children and Their Families
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Abd Elraheem Abd Elmonem, dentist, Cairo University
Other Study IDs: TDI
Record Dates: First submitted 2022-12-18; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Traumatic Dental Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of Impact of Complicated and Uncomplicated Traumatic Dental Injuries on Oral Health-Related Quality of Life in a Group of Preschool Children and Their Families.

DETAILED DESCRIPTION:
Statement of the problem Traumatic dental injury (TDI) is a current issue in public health (Milani et al, 2019). About one-third of children worldwide suffer from traumatic dental injuries (TDI), it has epidemiological significance. Throughout the child's growth and development, new and repetitive trauma may happen, influencing the dental, periodontal, bone, and soft tissue structures (Carneiro et al, 2020).

In young children, enamel fracture is the most frequent tooth injury, and this kind of trauma could go undetected by the child's parents, caregivers, or anybody else. The deciduous dentition has received a little amount of research on trauma (Carneiro et al, 2020).

Depending on the intensity of the consequences, dental trauma can have a significant impact on a child's life. It can cause discomfort and trouble chewing, as well as alter dento-facial aesthetics and, consequently, the person's ability to connect socially (Carneiro et al, 2020).

Systematic reviews have found that TDI affects pre-schoolers' oral health-related quality of life (OHRQoL). Children and their families suffer emotional and social consequences as a result (Antunes et al, 2020), (Zaror et al, 2018).

Risk factors, the impact of TDI, and the relation between TDI and socioeconomic status should all be considered (Antunes et al, 2020).

The purpose of this study is to assess the impact of dental trauma on children's and their families' oral health-related quality of life (OHRQoL), considering clinical and socioeconomic factors.

Rationale TDI cannot be anticipated and frequently requires emergency care due to its nature. Although it can happen at any age, the majority of TDI occurs in children. Literature reviews indicate that TDIs affect between one-third and one-fourth of kids in the primary dentition age range [(Jadav& Abbott, 2022), (Almeida et al, 2021)].

Due to the anatomical proximity of the germs of the permanent successors and the potential for adverse sequelae in both dentitions, TDI in the deciduous dentition requires extra care and attention. Therefore, the severity and extent of TDI can have an impact on the development of permanent successors as well as the prognosis of deciduous teeth (Antunes et al, 2020), (Andreasen et al, 2018).

Settings

• Location: preschool Nurseries in some rural areas in Elmaadi- Cairo.

* Methodology:
* Preschool children whose age ranged from 2 to yonger than 6 in some nurseries will be examined for traumatic dental injuries in anterior teeth.
* Examination will be performed in a room under natural light, with the help of wooden spatulas and gauze, by a single, trained and calibrated examiner.
* Type of tooth and the severity of TDI will be classified according to Glendor classification (Glendor et al, 1996) and will be recorded.
* The classification of Glenndor: Uncomplicated tooth injuries: in which the pulpal tissue are not exposed and/ or tooth is not dislocated. And Complicated tooth injuries: in which the pulpal tissue are exposed and/ or tooth is dislocated
* The author then will apply ECOHIS questionnaire on parents of children exposed to TDI after acceptance of informed consent.
* The questionnaire was developed by (Pahel et al, 2007)
* The questionnaire was then translated into Arabic and validated by (Nada Farsi et al, 2017).

ELIGIBILITY:
Inclusion Criteria:

* Children with traumatized primary teeth whose age ranges from 2<6, whose parents accept participation in study.

Exclusion Criteria:

* Children with mixed dentition.
* Children who presented absence of anterior teeth due to natural exfoliation
* Presence of crown defects not due to trauma.
* Children with previous orthodontic treatment or undergoing this treatment at the time of the study.
* Children with systemic or neuromotor diseases or had difficulties with communication.

Ages: 24 Months to 71 Months | Sex: All
Age Groups: Child
Study Population: Children with traumatized primary teeth whose age ranges from 2<6, whose parents accept participation in study.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Impact of Complicated and Uncomplicated Traumatic Dental Injuries on Oral Health-Related Quality of Life in a Group of Preschool Children and Their Families. | 12 months
  ECO HIS Questionnaire ECOHIS scores from 0 to 5
  Codes:
  0 = never
  1. = hardly ever
  2. = occasionally
  3. = often
  4. = very often
  5. = don't know

SECONDARY OUTCOMES:
Number of affected teeth in dentally traumatized preschool children | 12 months
  By clinical examination

REFERENCES:
- [Background] Antunes LAA, Milani AJ, Castilho T, Antunes LS. Impact of complicated and uncomplicated traumatic dental injuries on oral health-related quality of life of preschoolers and their family. Int J Burns Trauma. 2020 Aug 15;10(4):162-168. eCollection 2020. PMID 32934871
- [Background] Pahel BT, Rozier RG, Slade GD. Parental perceptions of children's oral health: the Early Childhood Oral Health Impact Scale (ECOHIS). Health Qual Life Outcomes. 2007 Jan 30;5:6. doi: 10.1186/1477-7525-5-6. PMID 17263880
- [Background] Glendor U, Halling A, Andersson L, Eilert-Petersson E. Incidence of traumatic tooth injuries in children and adolescents in the county of Vastmanland, Sweden. Swed Dent J. 1996;20(1-2):15-28. PMID 8738905